CLINICAL TRIAL: NCT06071637
Title: Low Power Laser Therapy As Prevention Of Oral Mucositis And Oropharyngeal Pain In Patients Undergoing Allogenetic Hematopoietic Stem Cell Transplantation.
Brief Title: Low Power Laser Therapy As Prevention Of Oral Mucositis And Oropharyngeal Pain In Patients Undergoing Allogenetic HSCT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 67172223.9.0000.5274
Record Dates: First submitted 2023-07-12; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-07

CONDITIONS: Hematopoietic Stem Cell Transplantation; Low-Level Light Therapy; Stomatitis
Keywords: Hematopoietic Stem Cell Transplantation; Low-Level Light Therapy; Stomatitis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Intervention Model Description: This is a phase III, double-blind, randomized intervention study that will use the low-power laser device to prevent oral mucositis and oropharyngeal pain in two protocols with different dosimetry (divided into Group A and Group B).
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization (simple) will be performed in permuted blocks using the REDCap® program, after inclusion in the study, by a member of the non-blinded team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - single emission (Active Comparator): The application will be carried out with the DMC device, with a power of 100mW, with a beam area of 0.09842 cm² in each optical fiber.
  Extraoral: A gallium and aluminum arsiade diode with emission of radiation in the infrared region of the electromagnetic spectrum (808 nm). An energy of 4J/point were determined, which will be applied punctually, with a distance between points of a maximum of 1cm, for 40s per point, totaling 9 points per region; Intraoral: An indium gallium aluminum phosphide diode with emission of radiation in the red region of the electromagnetic spectrum (660 nm). An energy of 1J/point were determined, which will be applied punctually, with a distance between points of a maximum of 1cm, for 10s per point, totaling 9 points per region .
  Interventions: Procedure: Double low-power laser therapy simultaneous applicated
- Group B - double emission (Experimental): The application will be carried out with the DMC device, with a power of 100mW, with a beam area of 0.09842 cm² in each optical fiber.
  Extraoral: An indium gallium aluminum phosphide diode and gallium aluminum arsiade with double radiation emission simultaneously in the red and infrared region of the electromagnetic spectrum (660 nm/808nm). An energy of 4J/point were determined, which will be applied punctually, with a maximum distance between points of 1cm, for 20s per point, totaling 9 points per region; Intraoral: An indium gallium aluminum phosphide diode and gallium aluminum arsiade with double radiation emission simultaneously in the red and infrared region of the electromagnetic spectrum (660nm/808nm). An energy of 1J / point (0.5J in the red and 0.5 in the infrared) were determined, which will be applied punctually, with a distance between points of no maximum 1cm, for 5s per point, totaling 9 points per region.
  Interventions: Procedure: Double low-power laser therapy simultaneous applicated

INTERVENTIONS:
Procedure: Double low-power laser therapy simultaneous applicated — Double low-power laser therapy, with simultaneous application of two wavelengths, red and infrared in in the mouth and neck

SUMMARY:
Objective: To compare the effects of two low-power laser therapy protocols (application of a wavelength in the mouth, red region and another in the neck infrared region X simultaneous dual application of two wavelengths, red and infrared region in the mouth and neck) in the prevention of oral mucositis and oropharyngeal pain, dysphagia, TPN and opioid use in patients undergoing HSCT allogenic.

Materials and methods: This is a phase III, double-blind, randomized study that will use LBP to prevent oral mucositis and oropharyngeal pain in two protocols with different dosimetry (divided into Group A and Group B). Patients will be included enrolled at the Bone Marrow Transplant Center - Cancer Hospital I - INCA, with indication of allogeneic HSCT, over 18 years old, able to cooperate with the treatment and perform the oral hygiene protocol, who present oral mucosa complete on the first day of conditioning (D-7) and who agree to participate in the study through the term of free and clarified informed consent. The randomization will be carried out in permuted blocks using the REDCap® program by a member of the non-blind team. In group A, extraoral applications will be carried out with the issuance of radiation in the infrared region of the electromagnetic spectrum (808nm) and intraorally in the red region of the electromagnetic spectrum (660nm). In group B, the extra applications and intraoral will be performed with simultaneous double radiation emission in the regions red and infrared of the electromagnetic spectrum (660nm/808nm). for both groups will use the device from DMC (São Carlos, São Paulo, Brazil), with a indium gallium aluminum phosphide (InGaAlP) and aluminum gallium arsiade diode (AlGaAs), with a power of 100mW and a beam area of 0.09842 cm². The LBP will be performed by a dental surgeon, on weekdays, starting on D-7 and end on the day of the "marrow take" (patient presents 500 neutrophils for three days consecutive). The region treated in extraoral applications will be the carotid triangle bilateral, bounded by the superior belly of the omohyoid, posterior belly of the digastric and by the anterior border of the sternocleidomastoid muscle; and intraorally, the mucous membranes right and left cheeks, lower and upper lips, upper and lower labial mucous membranes, right and left lateral borders of the tongue, lingual belly, buccal floor and soft palate. Patients will be evaluated daily (weekdays per week) for oral mucositis, pain in the oral cavity and oropharynx, dysphagia, use of total parenteral nutrition and opioids. Patients and dentists responsible for evaluating patients will be blinded to the study, that is, they will not know about the treatment that the patient will receive. The data from interest will be collected from the physical records and electronic systems of the institution, through standardized forms and will be included in REDCap®. Statistical analyzes will be carried out using the latest available version of the R software for Windows. It will be A descriptive analysis of the data found in the clinical, laboratory and sociodemographic data. To compare the incidence of mucositis, dysphagia, pain (treating the variables as dichotomous), the chi-square test of Pearson. Statistical analyzes will be performed using the latest available version of the R software for Windows. A descriptive analysis of the data found will be carried out in clinical examination, laboratory and sociodemographic data. To compare the incidence of mucositis, dysphagia, pain (treating the variables as dichotomous), the Pearson's chi-square test. Mucositis-free survival analyzes (any degree) and dysphagia (any degree) will be performed by the Kaplan-Meier method and the curves compared by log-rank test. The time interval between the start of conditioning and date of first grade ≥1 mucositis or dysphagia to date of the "marrow take" (500 neutrophils in the peripheral blood for three consecutive days). Participants without mucositis or dysphagia will be censored on the date of marrow collection. Tests of hypothesis with p-value < 0.05. The sample calculation predicted 82 patients, who will be evaluated by intention of treatment, counting with 10% loss to reach 37 patients in group A and 37 in group B. The estimate of the presence of oral mucositis grades 2, 3 and 4 in group A is 36.8% and in group B 10%. The estimate of the presence of dysphagia grades 3 and 4 (or pain in oropharynx grades 2 and 3) in group A is 80% and in group B 40%. the statistical test The two-tailed Z test with pooled variance was used, with a type 1 error of 0.05 and the error type 2 of 0.20. This research project was approved by the Research Ethics Committee responsible (CAAE 67172223.9.0000.5274, opinion No. 5.947.434) and will be conducted in a according to Resolution 466/12 of the National Health Council and the Good News Guide Clinical Practices.

DETAILED DESCRIPTION:
This is a phase III, double-blind, randomized study that will use low-power laser to prevent oral mucositis and oropharyngeal pain in two protocols with different dosimetry (divided into Group A and Group B).

The groups will be composed of patients evaluated in the Odontology Section of INCA, based on referrals from the Onco-Hematology team at the institution. After confirming the eligibility criteria, patients will be invited to participate in the research between the period of the pre-HSCT evaluation dental consultation and hospitalization for HSCT conditioning, and the TCLE will be applied according to the Good Clinical Practices Guide and the national ethical regulations. The TCLE must be applied before the D-7 or at the D-7 (beginning of conditioning). Randomization (simple) will be performed in permuted blocks using the REDCap® program, after inclusion in the study, by a member of the non-blinded team.

The pre-HSCT dental evaluation, according to the institutional routine, will consist of: intraoral physical examination performed by a dental surgeon (main researcher or another designated by him), radiographic examination (panoramic radiography) and pre-HSCT dental treatment (For example: resolution oral mucosa infections; removal of sources of trauma; scaling and root planing of teeth with 4-5mm periodontal pocket; restoration of minor carious lesions; adjustment or replacement of defective restorations; endodontic treatment of carious lesions with pulpal involvement, asymptomatic periapical lesion <1mm; extraction of teeth with abscesses, periapical lesion ≥1mm, or periodontal pocket ≥6mm, furcation lesion, mobility ≥2mm, partially erupted teeth, root remnants, intraosseous lesions, abnormalities such as root resorption; poorly fitting or removing prostheses adapted).

Participation in the study will end on the date of the "take" of the bone marrow. After that date, participants who present with oral mucositis will receive standard treatment according to the hospital's routine and will be followed up until the resolution of the event (More details in the section "Treatment of oral mucositis").

Prophylactic low-power laser therapy protocol

* The application of the low-power laser will be performed by a dental surgeon (main researcher or another designated by him), on weekdays, starting on the first day of conditioning (D-7) and ending on the day of "take the tooth". marrow" (patient presents 500 neutrophils for three consecutive days, the third consecutive day being considered the catch), which occurs on average between D+14 and D+21;
* In the extraoral application, the treated region will be the bilateral carotid triangle, limited by the superior belly of the omohyoid, posterior belly of the digastric and by the anterior margin of the sternocleidomastoid muscle.
* In the intraoral application, the treated regions of the oral mucosa will be: right and left buccal mucosa, lower and upper lip, upper and lower labial mucosa, right and left lateral edge of the tongue, lingual belly, buccal floor and soft palate.
* A power meter (Handheld Laser Power Meeter (RoHS) will be used weekly to assess the conditions of the device.
* The laser pointer will be disinfected with a 70% alcoholic solution, coated with a PVC film and disinfected with a 70% alcoholic solution. After the application of the laser, the PVC film will be removed and discarded, and then a new disinfection with 70% alcoholic solution of the device will be carried out;
* Patients and dentists will use protective eyewear, for individual use, with total light blocking during laser application, which will also be disinfected with a 70% alcoholic solution before and after use;
* The dentists responsible for applying the LBP will be previously trained;
* Patients and dentists responsible for evaluating patients will be blinded to the study, that is, they will not know what treatment the patient will receive. The mucositis evaluation step (blinded team) must occur before the laser application step (non-blinded team).

Oral hygiene protocol during HSCT Patients will be instructed to perform oral hygiene after all meals, solid or liquid, upon awakening and before going to sleep. In cases of exclusive use of TPN, patients will be instructed to brush their teeth three times a day. Oral hygiene will be carried out daily, from D-7 to taking the medulla, with a soft or extra soft brush and fluoride toothpaste.

Patients will be instructed to perform mouthwashes with a 0.12% chlorhexidine digluconate solution, a non-alcoholic solution, twice a day, from D-7 until the marrow takes hold.

The oral hygiene kit (toothbrush and toothpaste), 0.12% chlorhexidine digluconate solution will be routinely provided by the hospital to patients.

Signs of fungal infection will be considered, the characteristics of pseudomembranous and erythematous candidiasis described by Neville et al., (2016), where pseudomembranous candidiasis presents itself in the form of white, softened, detachable plaques, while the erythematous one is shown as red spots. From the diagnosis of fungal infection, patients will be treated according to the sector's routine and medical prescription.

Viral infections will be those that present themselves as multiple small and erythematous papules, which form groups of vesicles filled with liquid, which rupture, forming ulcers, which then form crusts within 2 days, thus characterizing a picture of herpes simplex. From the diagnosis of viral infection, patients will be treated according to the sector's routine and medical prescription.

Evaluation of oral mucositis The evaluation of oral mucositis will be carried out daily on weekdays, from D-7 until marrow attachment, by a blind sub-investigator, dental surgeon, previously designated by the main researcher, through intraoral physical examination. Weekly intraoral photographs will be taken from the first day of evaluation.

The WHO and OMAS scales will be used for the evaluation of oral mucositis. The WHO mucositis assessment scale consists of: grade 0, the patient does not have ulcers or erythema in the oral mucosa; grade 1, the patient does not have ulcers, but has erythema; grade 2, the patient has mouth ulcers, but manages to ingest solid foods and liquids; grade 3, the patient has mouth ulcers, but is able to ingest only liquid foods and in grade 4, the patient has mouth ulcers and is unable to ingest solid foods and liquids.

On the OMAS scale, the anatomical structures (upper and lower lips, right and left buccal mucosa, right and left tongue sides, dorsum and belly of the tongue, floor of the mouth, hard and soft palates) are scored according to the area of ulcerations and pseudomembranes, with the aid of a dental millimeter ruler (0: absent; 1: 1cm²; 2: 1 to 3cm² and 3: 3cm²) and erythema (0: absent; 1: Moderate and 2: Severe). Thus, the daily calculation of the sum of the weighted average of the ulcerated area and erythema intensity will be performed (MP=2.5 x [(∑ui : 3 x Nu )+ (∑ei: 2 x Ne)], where ∑ui= sum of ulcerated area, Nu= number of ulcerated areas, ∑ei= sum of erythema intensity and Ne= number of areas with erythema.

Treatment of oral mucositis From the diagnosis of oral mucositis, the patients will receive the therapeutic laser therapy protocol in the lesions, and will continue to receive the prophylactic in the other regions. The blind dentist (the evaluator) is the one who will define the moment of switching from the prophylactic to the therapeutic laser, according to the evaluation of the mucositis. The oral cavity assessment step (blinded team) precedes the laser application step (non-blinded team). The protocol will consist of daily applications (weekly working days), until the lesions are resolved, with an Indium-Gallium-Aluminum Phosphide (InGaAlP) laser diode, DMC, São Carlos, São Paulo, Brazil, with radiation emission in the region red light of the electromagnetic spectrum with 660nm, with power of 100mW, beam area of 0.09842 cm², 2J, 20.32J / cm².

Pain assessment The assessment of pain in the oral cavity will be performed daily, on weekdays, from D-7 until the marrow is taken, by a blind sub-investigator, dental surgeon, previously designated by the main researcher, according to the CTCAE scale v5.0 which classifies it as grade 1 (mild), grade 2 (moderate) with some limitation of daily activities and grade 3 (severe) with limitation of self-care in daily activities.

The assessment of pain in the oropharynx will be performed daily, on weekdays, from D-7 until the spinal cord is taken, by a blind sub-investigator, dental surgeon, previously designated by the main researcher, according to the CTCAE v5 scale .0, which classifies it as Grade 1 (mild pain), Grade 2 (moderate pain; altered oral intake; no use of narcotics; with topical analgesics started) and Grade 3 (severe pain; severely altered eating/swallowing; narcotics started; requires parenteral nutrition).

The CTCAE v5.0 scale will be associated with the pain scores of the Visual Analog Scale, where a value of 0 corresponds to the absence of pain and 10, the worst pain imaginable (Image 2). Will be considered: Absence of pain (zero); from 1 to 2 equivalent to a mild pain; from 3 to 7 moderate pain; and from 8 to 10, severe pain. Patients will be treated according to the sector's routine and medical prescription.

Dysphagia assessment Dysphagia assessment will be performed daily, on weekdays, from D-7 until marrow attachment, by a blind sub-investigator, dental surgeon, previously designated by the main researcher, according to the CTCAE v5.0 scale. They will be classified as: Absence of dysphagia (asymptomatic and able to eat a regular diet); Grade 1 (symptomatic, able to eat regular diet); Grade 2 (symptomatic with change in diet); Grade 3 (severely altered swallowing; TPN feeding); Grade 4 (Life-threatening consequences; urgent intervention indicated); and Grade 5 (death). Patients will be treated according to the sector's routine and medical prescription.

Evaluation of the use of total parenteral nutrition The presence or absence of TPN will be evaluated, and in cases where it is prescribed, the date of its onset until the marrow is taken will be recorded.

Evaluation of opioid use The presence or not of continuous prescription of opioids for the oral cavity/oropharynx will be evaluated, until the medulla takes hold. In cases where there is a prescription, the start date, substance and dosage will be recorded. The prescription will be carried out according to the sector's routine and medical prescription.

Data collect The data of interest will be collected from physical records and electronic systems of the institution, through standardized forms and will be included in REDCap®, an electronic data collection system, in customized forms for this research project.

In the clinical evaluation form 1 (Appendix 1) data will be recorded regarding age (in years), date of birth, sex (female and male), underlying disease, associated comorbidities, date of hospitalization for HSCT, conditioning protocol , conditioning start date, HSCT date, marrow take date, length of stay during HSCT (considering the start of conditioning) and drugs prescribed for GVHD prophylaxis.

In the clinical evaluation form 2 (Appendix 2), data referring to the mucositis evaluations by the WHO and OMAS, visual analogue scale for pain in the oral cavity and oropharynx, CTCAE v5.0 scale for pain in the oral cavity, oropharynx and dysphagia, TPN and use of opioids.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for allogeneic HSCT;
* Patients over 18 years old;
* Patients with intact oral mucosa on the first day of conditioning (D-7);
* Patients able to cooperate with treatment;
* Patients capable of performing the oral hygiene protocol;
* Patients who agreed to participate in the study through the informed consent form (TCLE) in accordance with Resolution 466/12 of the National Health Council.

Exclusion Criteria:

* Patients who are receiving medication for the treatment and/or prevention of mucositis;
* Patients who were not previously evaluated and released by INCA's Dentistry section team

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Prevention of oral mucositis according to WHO and OMAS scale | During the period of hospitalization due to HSCT, approximately 21 to 28 days
Prevention of oropharyngeal pain according to the CTCAE v5.0 and the Visual Analog Scale | During the period of hospitalization due to HSCT, approximately 21 to 28 days
Prevention of dysphagia according to the CTCAE v5.0 scale | During the period of hospitalization due to HSCT, approximately 21 to 28 days
Prevention of the need for total parenteral nutrition | During the period of hospitalization due to HSCT, approximately 21 to 28 days
Prevention of the need for opioid use | During the period of hospitalization due to HSCT, approximately 21 to 28 days

SECONDARY OUTCOMES:
Association between the incidence of oral mucositis (any degree) and the prophylactic laser therapy protocol used | During the period of hospitalization due to HSCT, approximately 21 to 28 days
Association between the incidence of pain in the oral cavity and oropharynx (any degree) and the prophylactic laser therapy protocol used | During the period of hospitalization due to HSCT, approximately 21 to 28 days
Association between the incidence of dysphagia (any degree) and the prophylactic laser therapy protocol used | During the period of hospitalization due to HSCT, approximately 21 to 28 days
Association between oral mucositis-free survival (any grade) and the prophylactic laser therapy protocol used | During the period of hospitalization due to HSCT, approximately 21 to 28 days
Association between dysphagia-free survival (any degree) and the prophylactic laser therapy protocol used | During the period of hospitalization due to HSCT, approximately 21 to 28 days
Association between the use of Total Parenteral Nutrition (TPN) and the prophylactic laser therapy protocol used | During the period of hospitalization due to HSCT, approximately 21 to 28 days
Association between the use of opioids (prescribed for pain in the oral cavity/oropharynx) and the prophylactic laser therapy protocol used | During the period of hospitalization due to HSCT, approximately 21 to 28 days

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Instituto Nacional de Cancer, Rio de Janeiro, Rio de Janeiro
  - Instituto Nacional de Cancer, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No
Data will be relased after the study is completd.

REFERENCES:
- [Background] Adnan A, Yaroslavsky AN, Carroll JD, Selting W, Juliano AF, London WB, Sonis ST, Duncan CN, Treister NS. The Path to an Evidence-Based Treatment Protocol for Extraoral Photobiomodulation Therapy for the Prevention of Oral Mucositis. Front Oral Health. 2021 Jul 16;2:689386. doi: 10.3389/froh.2021.689386. eCollection 2021. PMID 35048034
- [Background] ALVES, L. D. B. et al. Strategies for the dentist management of cancer patients: narrative literature review. Journal of Cancer Prevention & Current Research Review, v. 12, n. 4, p. 111-121, 2021.
- [Background] ANTUNES, H. S. et al. Como o cirurgião dentista deve atender o paciente oncológico?Rev. Int. Estomatol, 2004.
- [Background] Antunes HS, de Azevedo AM, da Silva Bouzas LF, Adao CA, Pinheiro CT, Mayhe R, Pinheiro LH, Azevedo R, D'Aiuto de Matos V, Rodrigues PC, Small IA, Zangaro RA, Ferreira CG. Low-power laser in the prevention of induced oral mucositis in bone marrow transplantation patients: a randomized trial. Blood. 2007 Mar 1;109(5):2250-5. doi: 10.1182/blood-2006-07-035022. Epub 2006 Oct 19. PMID 17053058
- [Background] Armitage JO. Bone marrow transplantation. N Engl J Med. 1994 Mar 24;330(12):827-38. doi: 10.1056/NEJM199403243301206. No abstract available. PMID 8114836
- [Background] ASSOCIAÇÃO DA MEDULA ÓSSEA DO ESTADO DE SÃO PAULO. Mapa do Transplante de Medula Óssea. Disponível em: <https://www.rowconsultoria.com.br/ameo/dashp.aspx>. Acesso em: 27 set. 2022.
- [Background] Balassa K, Danby R, Rocha V. Haematopoietic stem cell transplants: principles and indications. Br J Hosp Med (Lond). 2019 Jan 2;80(1):33-39. doi: 10.12968/hmed.2019.80.1.33. PMID 30592675
- [Background] de Castro CG Jr, Gregianin LJ, Brunetto AL. [Bone marrow transplantation and cord blood transplantation in children]. J Pediatr (Rio J). 2001 Sep-Oct;77(5):345-60. doi: 10.2223/jped.275. Portuguese. PMID 14647838
- [Background] Chaudhry HM, Bruce AJ, Wolf RC, Litzow MR, Hogan WJ, Patnaik MS, Kremers WK, Phillips GL, Hashmi SK. The Incidence and Severity of Oral Mucositis among Allogeneic Hematopoietic Stem Cell Transplantation Patients: A Systematic Review. Biol Blood Marrow Transplant. 2016 Apr;22(4):605-616. doi: 10.1016/j.bbmt.2015.09.014. Epub 2015 Sep 26. PMID 26409924
- [Background] Copelan EA. Hematopoietic stem-cell transplantation. N Engl J Med. 2006 Apr 27;354(17):1813-26. doi: 10.1056/NEJMra052638. No abstract available. PMID 16641398
- [Background] Corazza AV, Jorge J, Kurachi C, Bagnato VS. Photobiomodulation on the angiogenesis of skin wounds in rats using different light sources. Photomed Laser Surg. 2007 Apr;25(2):102-6. doi: 10.1089/pho.2006.2011. PMID 17508845
- [Background] Elad S, Raber-Durlacher JE, Brennan MT, Saunders DP, Mank AP, Zadik Y, Quinn B, Epstein JB, Blijlevens NM, Waltimo T, Passweg JR, Correa ME, Dahllof G, Garming-Legert KU, Logan RM, Potting CM, Shapira MY, Soga Y, Stringer J, Stokman MA, Vokurka S, Wallhult E, Yarom N, Jensen SB. Basic oral care for hematology-oncology patients and hematopoietic stem cell transplantation recipients: a position paper from the joint task force of the Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO) and the European Society for Blood and Marrow Transplantation (EBMT). Support Care Cancer. 2015 Jan;23(1):223-36. doi: 10.1007/s00520-014-2378-x. Epub 2014 Sep 5. PMID 25189149
- [Background] Elad S, Cheng KKF, Lalla RV, Yarom N, Hong C, Logan RM, Bowen J, Gibson R, Saunders DP, Zadik Y, Ariyawardana A, Correa ME, Ranna V, Bossi P; Mucositis Guidelines Leadership Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer. 2020 Oct 1;126(19):4423-4431. doi: 10.1002/cncr.33100. Epub 2020 Jul 28. PMID 32786044
- [Background] Ferreira B, da Motta Silveira FM, de Orange FA. Low-level laser therapy prevents severe oral mucositis in patients submitted to hematopoietic stem cell transplantation: a randomized clinical trial. Support Care Cancer. 2016 Mar;24(3):1035-42. doi: 10.1007/s00520-015-2881-8. Epub 2015 Aug 7. PMID 26248655
- [Background] Ferreira E, Dulley FL, Morsoletto F, Neto JZ, Pasquini R. Bone marrow transplantation in Brazil. Hum Immunol. 1985 Nov;14(3):324-32. doi: 10.1016/0198-8859(85)90240-x. PMID 3902750
- [Background] Franca CM, Franca CM, Nunez SC, Prates RA, Noborikawa E, Faria MR, Ribeiro MS. Low-intensity red laser on the prevention and treatment of induced-oral mucositis in hamsters. J Photochem Photobiol B. 2009 Jan 9;94(1):25-31. doi: 10.1016/j.jphotobiol.2008.09.006. Epub 2008 Sep 30. PMID 18976931
- [Background] Hodgson BD, Margolis DM, Salzman DE, Eastwood D, Tarima S, Williams LD, Sande JE, Vaughan WP, Whelan HT. Amelioration of oral mucositis pain by NASA near-infrared light-emitting diodes in bone marrow transplant patients. Support Care Cancer. 2012 Jul;20(7):1405-15. doi: 10.1007/s00520-011-1223-8. Epub 2011 Jul 3. PMID 21725826
- [Background] INSTITUTO NACIONAL DE CÂNCER. Cuidados paliativos oncológicos. Rio de Janeiro: Ministério da Saúde do Brasil, 2001. v. 22
- [Background] INSTITUTO NACIONAL DE CÂNCER JOSÉ ALENCAR GOMES DA SILVA. Estimativa 2023: incidêcia de câncer no Brasil. Disponível em: <https://www.gov.br/inca/pt-br/assuntos/cancer/numeros/estimativa/estado-capital/brasil>. Acesso em: 25 nov. 2022.
- [Background] Karu TI, Pyatibrat LV, Kalendo GS. Photobiological modulation of cell attachment via cytochrome c oxidase. Photochem Photobiol Sci. 2004 Feb;3(2):211-6. doi: 10.1039/b306126d. Epub 2003 Nov 12. PMID 14872239
- [Background] Khaddour K, Hana CK, Mewawalla P. Hematopoietic Stem Cell Transplantation. 2023 May 6. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK536951/ PMID 30725636
- [Background] Khouri VY, Stracieri AB, Rodrigues MC, Moraes DA, Pieroni F, Simoes BP, Voltarelli JC. Use of therapeutic laser for prevention and treatment of oral mucositis. Braz Dent J. 2009;20(3):215-20. doi: 10.1590/s0103-64402009000300008. PMID 19784467
- [Background] KRESLAVSKI, V. D. et al. Red and near infra-red signaling: Hypothesis and perspectives. Journal of Photochemistry and Photobiology C: Photochemistry Reviews, v. 13, n. 3, p. 190-203, 2012.
- [Background] Lalla RV, Bowen J, Barasch A, Elting L, Epstein J, Keefe DM, McGuire DB, Migliorati C, Nicolatou-Galitis O, Peterson DE, Raber-Durlacher JE, Sonis ST, Elad S; Mucositis Guidelines Leadership Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer. 2014 May 15;120(10):1453-61. doi: 10.1002/cncr.28592. Epub 2014 Feb 25. PMID 24615748
- [Background] Magedanz L, Leal JVO, Santos BLD, Brito ES, Saavedra PAE, Soares LSDS, D'Oliveira LDCL, Galato D. [Hematopoietic stem-cell transplants in Brazil: inequities in the distribution in Brazilian territory, 2001 to 2020]. Cien Saude Colet. 2022 Aug;27(8):3239-3247. doi: 10.1590/1413-81232022278.03142022. Epub 2022 Apr 16. Portuguese. PMID 35894334
- [Background] MENEZES, A. C. et al. Abordagem clínica e terapêutica da mucosite oral induzida por radioterapia e quimioterapia em pacientes com câncer. Revistas, v. 71, n. 1, p. 35, 2014.
- [Background] Nakagaki M, Kennedy GA, Gavin NC, Clavarino A, Whitfield K. The incidence of severe oral mucositis in patients undergoing different conditioning regimens in haematopoietic stem cell transplantation. Support Care Cancer. 2022 Nov;30(11):9141-9149. doi: 10.1007/s00520-022-07328-4. Epub 2022 Aug 26. PMID 36008731
- [Background] NATIONAL CANCER INSTITUTE OF USA. Common Terminology Criteria for Adverse Events, Version 5.0. In: Definitions. [s.l.] Qeios, 2017.
- [Background] NEVILLE, B. W. et al. Patologia oral e maxilofacial. 4. ed. Rio de Janeiro: Elsevier, 2016.
- [Background] Ramos-Pinto MB, de Lima Gusmao TP, Schmidt-Filho J, Jaguar GC, Martins MD, Alves FA. Intraoral versus extraoral photobiomodulation therapy in the prevention of oral mucositis in HSCT patients: a randomized, single-blind, controlled clinical trial. Support Care Cancer. 2021 Nov;29(11):6495-6503. doi: 10.1007/s00520-021-06228-3. Epub 2021 Apr 27. PMID 33905011
- [Background] SANTOS, P. S. D. S. et al. Mucosite oral: perspectivas atuais na prevenção e tratamento. Revista Gaúcha de Odontologia, v. 57, n. 3, p. 339-344, 2009.
- [Background] Schubert MM, Eduardo FP, Guthrie KA, Franquin JC, Bensadoun RJ, Migliorati CA, Lloid CM, Eduardo CP, Walter NF, Marques MM, Hamdi M. A phase III randomized double-blind placebo-controlled clinical trial to determine the efficacy of low level laser therapy for the prevention of oral mucositis in patients undergoing hematopoietic cell transplantation. Support Care Cancer. 2007 Oct;15(10):1145-54. doi: 10.1007/s00520-007-0238-7. Epub 2007 Mar 29. PMID 17393191
- [Background] SCHUSTER, A.; BASSANI, B.; FARIAS, E. Epidemiologia dos transplantes de medula óssea entre 2010 e 2019 no Brasil. Hematology, Transfusion and Cell Therapy, v. 43, p. S258, out. 2021.
- [Background] Shouval R, Kouniavski E, Fein J, Danylesko I, Shem-Tov N, Geva M, Yerushalmi R, Shimoni A, Nagler A. Risk factors and implications of oral mucositis in recipients of allogeneic hematopoietic stem cell transplantation. Eur J Haematol. 2019 Oct;103(4):402-409. doi: 10.1111/ejh.13299. Epub 2019 Aug 12. PMID 31332836
- [Background] Silva GB, Mendonca EF, Bariani C, Antunes HS, Silva MA. The prevention of induced oral mucositis with low-level laser therapy in bone marrow transplantation patients: a randomized clinical trial. Photomed Laser Surg. 2011 Jan;29(1):27-31. doi: 10.1089/pho.2009.2699. Epub 2010 Oct 22. PMID 20969443
- [Background] Silva LC, Sacono NT, Freire Mdo C, Costa LR, Batista AC, Silva GB. The Impact of Low-Level Laser Therapy on Oral Mucositis and Quality of Life in Patients Undergoing Hematopoietic Stem Cell Transplantation Using the Oral Health Impact Profile and the Functional Assessment of Cancer Therapy-Bone Marrow Transplantation Questionnaires. Photomed Laser Surg. 2015 Jul;33(7):357-63. doi: 10.1089/pho.2015.3911. PMID 26154723
- [Background] Sonis ST, Eilers JP, Epstein JB, LeVeque FG, Liggett WH Jr, Mulagha MT, Peterson DE, Rose AH, Schubert MM, Spijkervet FK, Wittes JP. Validation of a new scoring system for the assessment of clinical trial research of oral mucositis induced by radiation or chemotherapy. Mucositis Study Group. Cancer. 1999 May 15;85(10):2103-13. doi: 10.1002/(sici)1097-0142(19990515)85:103.0.co;2-0. PMID 10326686
- [Background] Sonis ST. The pathobiology of mucositis. Nat Rev Cancer. 2004 Apr;4(4):277-84. doi: 10.1038/nrc1318. No abstract available. PMID 15057287
- [Background] Soto M, Lalla RV, Gouveia RV, Zecchin VG, Seber A, Lopes NN. Pilot study on the efficacy of combined intraoral and extraoral low-level laser therapy for prevention of oral mucositis in pediatric patients undergoing hematopoietic stem cell transplantation. Photomed Laser Surg. 2015 Nov;33(11):540-6. doi: 10.1089/pho.2015.3954. Epub 2015 Oct 26. PMID 26501372
- [Background] Whelan HT, Connelly JF, Hodgson BD, Barbeau L, Post AC, Bullard G, Buchmann EV, Kane M, Whelan NT, Warwick A, Margolis D. NASA light-emitting diodes for the prevention of oral mucositis in pediatric bone marrow transplant patients. J Clin Laser Med Surg. 2002 Dec;20(6):319-24. doi: 10.1089/104454702320901107. PMID 12513918
- [Background] WORLD HEALTH ORGANIZATION /WHO. WHO handbook for reporting results of cancer treatmentInternational Journal of Radiation Biology, 1979.
- [Background] Zadik Y, Arany PR, Fregnani ER, Bossi P, Antunes HS, Bensadoun RJ, Gueiros LA, Majorana A, Nair RG, Ranna V, Tissing WJE, Vaddi A, Lubart R, Migliorati CA, Lalla RV, Cheng KKF, Elad S; Mucositis Study Group of the Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO). Systematic review of photobiomodulation for the management of oral mucositis in cancer patients and clinical practice guidelines. Support Care Cancer. 2019 Oct;27(10):3969-3983. doi: 10.1007/s00520-019-04890-2. Epub 2019 Jul 8. PMID 31286228